CLINICAL TRIAL: NCT01080846
Title: Assessment of Fever After Misoprostol Administration for the Treatment of Primary Postpartum Hemorrhage
Brief Title: Fever After Misoprostol Administration for the Treatment of Primary Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Liverpool (Other)
Responsible Party: Jill Durocher, Program Associate, Gynuity Health Projects
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.4.6
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Postpartum Hemorrhage
Keywords: Primary postpartum hemorrhage; PPH; uterine atony; high fever; hyperpyrexia
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Inertia; Hyperthermia | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 600 mcg of sublingual misoprostol (Experimental)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 600 mcg of sublingual misoprostol

SUMMARY:
This study will evaluate side effects after sublingual misoprostol (600 mcg) as a first-line treatment for primary postpartum hemorrhage (PPH) due to suspected uterine atony.

DETAILED DESCRIPTION:
The study purpose is to confirm whether a lower, 600 mcg dose of sublingual misoprostol will reduce the incidence of elevated body temperature (≥40°C) associated with misoprostol. The study will compare the incidence of high fevers following treatment with 600 mcg sublingual misoprostol to previously documented rates using 800 mcg sublingual misoprostol. An additional line of research is to investigate whether some women are more susceptible to experiencing high fevers following misoprostol administration, and whether genetic factors are responsible for misoprostol-induced fevers.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent
* Vaginal delivery
* Postpartum hemorrhage due to suspected uterine atony
* Oxytocin given during 3rd stage of labor

Exclusion Criteria:

* Known allergy to prostaglandins or misoprostol
* Underwent cesarean section
* Postpartum hemorrhage NOT due to suspected uterine atony
* Oxytocin NOT given during 3rd stage of labor
* Severe ill health
* Unable to give informed consent

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Rate of fever above 40.0 degrees centigrade | Body temperature measured at 60 minutes and 90 minutes post-treatment with misoprostol for PPH
  % of women with body temperature measures ≥40°C

SECONDARY OUTCOMES:
Side effect profile of misoprostol for PPH treatment | Side effects observed for 3 hours post-treatment with misoprostol for PPH
  % of women experiencing any shivering and any fever or any other side effect
Acceptability of side effect profile among women | Women interviewed prior to hospital discharge about acceptability of side effects (24 hours postpartum)
  % of women who rate side effects as acceptable, neutral, unacceptable, don't know

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Andrew Weeks, MD, Principal Investigator — The University of Liverpool; Wilfrido Leon, MD, Principal Investigator — HOSPITAL GINECO OBSTETRICO ISIDRO AYORA; Gustavo Barrera, MD, Principal Investigator — HOSPITAL GINECO OBSTETRICO ISIDRO AYORA; Jill Durocher, Principal Investigator — Gynuity Health Projects
Locations (1):
- Hospital Gineco Obstetrico Isidro Ayora, Quito, Pichincha, Ecuador

REFERENCES:
- [Background] Winikoff B, Dabash R, Durocher J, Darwish E, Nguyen TN, Leon W, Raghavan S, Medhat I, Huynh TK, Barrera G, Blum J. Treatment of post-partum haemorrhage with sublingual misoprostol versus oxytocin in women not exposed to oxytocin during labour: a double-blind, randomised, non-inferiority trial. Lancet. 2010 Jan 16;375(9710):210-6. doi: 10.1016/S0140-6736(09)61924-3. Epub 2010 Jan 6. PMID 20060161
- [Background] Blum J, Winikoff B, Raghavan S, Dabash R, Ramadan MC, Dilbaz B, Dao B, Durocher J, Yalvac S, Diop A, Dzuba IG, Ngoc NT. Treatment of post-partum haemorrhage with sublingual misoprostol versus oxytocin in women receiving prophylactic oxytocin: a double-blind, randomised, non-inferiority trial. Lancet. 2010 Jan 16;375(9710):217-23. doi: 10.1016/S0140-6736(09)61923-1. Epub 2010 Jan 6. PMID 20060162
- [Derived] Leon W, Durocher J, Barrera G, Pinto E, Winikoff B. Dose and side effects of sublingual misoprostol for treatment of postpartum hemorrhage: what difference do they make? BMC Pregnancy Childbirth. 2012 Jul 7;12:65. doi: 10.1186/1471-2393-12-65. PMID 22769055
- See also: Gynuity Health Projects — http://www.gynuity.org